CLINICAL TRIAL: NCT04566029
Title: Analysis of the Evolution of Proteomic Profiles of Intestinal Microbiota in Patients With Locally Advanced or Metastatic Urothelial Carcinomas According to Their Response to Immunotherapy (Responders vs. Non-responders) : A Prospective Pilot Study
Brief Title: Evolution of Proteomic Profiles of Intestinal Microbiota in Patients With Locally Advanced or Metastatic Urothelial Carcinomas
Acronym: AMI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: European Georges Pompidou Hospital (Other); ICM Montpellier (Unknown); IUCT Oncopole (Toulouse) (Unknown); Institut de cancérologie Strasbourg Europe (Other); Institut de Cancérologie Lucien Neuwirth (Saint Etienne) (Unknown); ICO - SITE Paul Papin (Unknown); Centre Antoine Lacassagne (Other); Institut Bergonié (Other); Tenon Hospital, Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO2019_2; 2020-A01224-35 (Other: ANSM)
Record Dates: First submitted 2020-08-06; First posted 2020-09-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Hematologic Tests; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients who have been responding to treatment for a long time
  Interventions: Biological: Blood test; Biological: Stool sample; Other: Questionnaires
- Controls: Patients who do not respond to treatment
  Interventions: Biological: Blood test; Biological: Stool sample; Other: Questionnaires

INTERVENTIONS:
Biological: Blood test — The patients' blood will be collected in four 5mL heparinized tubes
Biological: Stool sample — The patients' stools will be collected at home
Other: Questionnaires — At each visit, the following questionnaires will be collected: QLQ-C30 and EQ5D-5L Appendix 16.2 and PRO CTCAE

SUMMARY:
Immunotherapy has become an essential therapeutic weapon against many cancers. Control point inhibitors (CPI, PD-1/PD-L1) have shown efficacy in the therapeutic management of tumors in the bladder in progression after administering platinum derivatives. But only 20% of patients get any clinical benefit from these heavy treatments in the long term.

Treating metastatic patients without distinction means taking a considerable risk of toxicity and generates major costs. It is therefore urgent and important to exceed the current criteria for using immunotherapy. Recent studies have shown the interest of studying intestinal microbiota as a marker of the efficacy of immunotherapy.

The investigators hypothesized that the proteomic signature of the intestinal microbiota in patients with locally advanced or metastatic urothelial carcinomas who responded to immunotherapies was special, and has very different characteristics from that of patients with the same pathology who do not respond to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

For the "controls" group:

* Patients undergoing treatment for a locally advanced or metastatic urothelial tumor
* Patients who have been on immunotherapy and 2nd-line monotherapy treatment for at least 6 months for a non-operable disease
* Patients whose immunotherapy has been interrupted due to progression of the disease

For the "cases" group:

* patients being treated in the context of a temporary authorization for use delivered for atezolizumab for the management of locally advanced or metastatic urothelial carcinomas following treatment based on platinum salts and still on treatment or patients being treated with pembrolizumab in the context of a donation for compassionate reasons (and still on treatment).

Exclusion Criteria:

* Patients who do not speak or read the French language.
* Patients in an exclusion period determined by another study.
* Patients under legal guardianship or curatorship.
* Patients for whom it is impossible to give clear information to.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are affiliated to or covered by a health insurance scheme. All patients over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Stool sample collected from patients in the "cases" group | 24 hours before the patient's follow-up visit at 1 month +/- 7 days
  Quantification of bacterial proteins as a reflection of the intestinal microbiota and human proteins in the patient's stools. These will be analyzed from 50mg of stools via mass spectrometry (ESI-Q combined with the Ultimate 3000 Nano liquid chromatography system, ThermoFisher Scientific).
Stool sample collected from patients in the "controls" group | 24 hours before the patient's follow-up visit at 1 month +/- 7 days
  Quantification of bacterial proteins as a reflection of the intestinal microbiota and human proteins in the patient's stools.These will be analyzed from 50mg of stools via mass spectrometry (ESI-Q combined with the Ultimate 3000 Nano liquid chromatography system, ThermoFisher Scientific).

SECONDARY OUTCOMES:
Immune system markers in patients with locally advanced or metastatic urothelial carcinomas in "cases" group patients. | At the follow-up visit, 1 month +/- 7 days after inclusion
  For each patient in the "cases" group, blood will be collected in four heparinized tubes and the immune populations will be studied via mass spectrometry (CyTOF/Helios). The frequency of the subpopulations thus determined will be compared between the two groups of patients (responders vs non responders) in order to identify those populations which are significantly different.
Immune system markers in patients with locally advanced or metastatic urothelial carcinomas in "controls" group patients. | At the follow-up visit, 1 month +/- 7 days after inclusion
  For each patient in the "controls" group, blood will be collected in four heparinized tubes and the immune populations will be studied via mass spectrometry (CyTOF/Helios). The frequency of the subpopulations thus determined will be compared between the two groups of patients (responders vs non responders) in order to identify those populations which are significantly different.
Evolution over time in the quality of life of patients in the "cases" group - EORTC QLQ-C30 | At the inclusion visit on Day 0
  The quality of life will be evaluated via the EORTC QLQ-C30 questionnaire. The quality of life questionnaire designed by the European Organisation for Research and Treatment of Cancer known as EORTC QLQ-C30 is for all cancer patients, whatever the location of their cancer. It consists of 30 items grouped together into 15 dimensions. There are 4 possible answers to the first 28 items and 7 possible answers to the last 2 questions. The answers take the form of a Lickert scale.
Evolution over time in the quality of life of patients in the "cases" group - EORTC QLQ-C30 | At the follow-up visit, 1 month +/- 7 days after inclusion
  The quality of life will be evaluated via the EORTC QLQ-C30 questionnaire. The quality of life questionnaire designed by the European Organisation for Research and Treatment of Cancer known as EORTC QLQ-C30 is for all cancer patients, whatever the location of their cancer. It consists of 30 items grouped together into 15 dimensions. There are 4 possible answers to the first 28 items and 7 possible answers to the last 2 questions. The answers take the form of a Lickert scale.
Evolution over time in the quality of life of patients in the "cases" group - EORTC QLQ-C30 | At the end of study visit, 2 months +/- 15 days after inclusion
  The quality of life will be evaluated via the EORTC QLQ-C30 questionnaire. The quality of life questionnaire designed by the European Organisation for Research and Treatment of Cancer known as EORTC QLQ-C30 is for all cancer patients, whatever the location of their cancer. It consists of 30 items grouped together into 15 dimensions. There are 4 possible answers to the first 28 items and 7 possible answers to the last 2 questions. The answers take the form of a Lickert scale.
Evolution over time in the quality of life of patients in the "controls" group - EORTC QLQ-C30 | At the inclusion visit on Day 0
  The quality of life will be evaluated via the EORTC QLQ-C30 questionnaire. The quality of life questionnaire designed by the European Organisation for Research and Treatment of Cancer known as EORTC QLQ-C30 is for all cancer patients, whatever the location of their cancer. It consists of 30 items grouped together into 15 dimensions. There are 4 possible answers to the first 28 items and 7 possible answers to the last 2 questions. The answers take the form of a Lickert scale.
Evolution over time in the quality of life of patients in the "controls" group - EORTC QLQ-C30 | At the follow-up visit, 1 month +/- 7 days after inclusion
  The quality of life will be evaluated via the EORTC QLQ-C30 questionnaire. The quality of life questionnaire designed by the European Organisation for Research and Treatment of Cancer known as EORTC QLQ-C30 is for all cancer patients, whatever the location of their cancer. It consists of 30 items grouped together into 15 dimensions. There are 4 possible answers to the first 28 items and 7 possible answers to the last 2 questions. The answers take the form of a Lickert scale.
Evolution over time in the quality of life of patients in the "controls" group - EORTC QLQ-C30 | At the end of study visit, 2 months +/- 15 days after inclusion
  The quality of life will be evaluated via the EORTC QLQ-C30 questionnaire. The quality of life questionnaire designed by the European Organisation for Research and Treatment of Cancer known as EORTC QLQ-C30 is for all cancer patients, whatever the location of their cancer. It consists of 30 items grouped together into 15 dimensions. There are 4 possible answers to the first 28 items and 7 possible answers to the last 2 questions. The answers take the form of a Lickert scale.
Evolution over time in the quality of life of patients in the "cases" group - EQ5D-5L | At the inclusion visit on Day 0
  The EQ-5D (EuroQoL -5 Dimension) self-report questionnaire will be used to measure the quality of life under various health conditions and treatments according to 5 dimensions: mobility, personal autonomy, everyday living activities, pain/discomfort and anxiety/depression. There are 3 versions of this questionnaire: EQ-5D-3L with 3 levels of severity for each dimension, EQ-5D-5L with 5 levels of severity for each dimension and EQ-5D-Y which is the children's version. Each version is available in several languages. The questionnaire has 2 pages : page one with 5 items representing the 5 dimensions and page two with a visual analogue scale graded from 0 to 100 with 100 as the best possible state of health. For each dimension the patient must indicate what condition he/she is in. When all the answers are combined, a 5-figure number is obtained, indicating the patient's health condition. For example, the number 11111 shows that there are no problems in any of the 5 dimensions.
Evolution over time in the quality of life of patients in the "cases" group - EQ5D-5L | At the follow-up visit, 1 month +/- 7 days after inclusion
  The EQ-5D (EuroQoL -5 Dimension) self-report questionnaire will be used to measure the quality of life under various health conditions and treatments according to 5 dimensions: mobility, personal autonomy, everyday living activities, pain/discomfort and anxiety/depression. There are 3 versions of this questionnaire: EQ-5D-3L with 3 levels of severity for each dimension, EQ-5D-5L with 5 levels of severity for each dimension and EQ-5D-Y which is the children's version. Each version is available in several languages. The questionnaire has 2 pages : page one with 5 items representing the 5 dimensions and page two with a visual analogue scale graded from 0 to 100 with 100 as the best possible state of health. For each dimension the patient must indicate what condition he/she is in. When all the answers are combined, a 5-figure number is obtained, indicating the patient's health condition. For example, the number 11111 shows that there are no problems in any of the 5 dimensions.
Evolution over time in the quality of life of patients in the "cases" group - EQ5D-5L | At the end of study visit, 2 months +/- 15 days after inclusion
  The EQ-5D (EuroQoL -5 Dimension) self-report questionnaire will be used to measure the quality of life under various health conditions and treatments according to 5 dimensions: mobility, personal autonomy, everyday living activities, pain/discomfort and anxiety/depression. There are 3 versions of this questionnaire: EQ-5D-3L with 3 levels of severity for each dimension, EQ-5D-5L with 5 levels of severity for each dimension and EQ-5D-Y which is the children's version. Each version is available in several languages. The questionnaire has 2 pages : page one with 5 items representing the 5 dimensions and page two with a visual analogue scale graded from 0 to 100 with 100 as the best possible state of health. For each dimension the patient must indicate what condition he/she is in. When all the answers are combined, a 5-figure number is obtained, indicating the patient's health condition. For example, the number 11111 shows that there are no problems in any of the 5 dimensions.
Evolution over time in the quality of life of patients in the "controls" group - EQ5D-5L | At the inclusion visit on Day 0
  The EQ-5D (EuroQoL -5 Dimension) self-report questionnaire will be used to measure the quality of life under various health conditions and treatments according to 5 dimensions: mobility, personal autonomy, everyday living activities, pain/discomfort and anxiety/depression. There are 3 versions of this questionnaire: EQ-5D-3L with 3 levels of severity for each dimension, EQ-5D-5L with 5 levels of severity for each dimension and EQ-5D-Y which is the children's version. Each version is available in several languages. The questionnaire has 2 pages : page one with 5 items representing the 5 dimensions and page two with a visual analogue scale graded from 0 to 100 with 100 as the best possible state of health. For each dimension the patient must indicate what condition he/she is in. When all the answers are combined, a 5-figure number is obtained, indicating the patient's health condition. For example, the number 11111 shows that there are no problems in any of the 5 dimensions.
Evolution over time in the quality of life of patients in the "controls" group - EQ5D-5L | At the follow-up visit, 1 month +/- 7 days after inclusion
  The EQ-5D (EuroQoL -5 Dimension) self-report questionnaire will be used to measure the quality of life under various health conditions and treatments according to 5 dimensions: mobility, personal autonomy, everyday living activities, pain/discomfort and anxiety/depression. There are 3 versions of this questionnaire: EQ-5D-3L with 3 levels of severity for each dimension, EQ-5D-5L with 5 levels of severity for each dimension and EQ-5D-Y which is the children's version. Each version is available in several languages. The questionnaire has 2 pages : page one with 5 items representing the 5 dimensions and page two with a visual analogue scale graded from 0 to 100 with 100 as the best possible state of health. For each dimension the patient must indicate what condition he/she is in. When all the answers are combined, a 5-figure number is obtained, indicating the patient's health condition. For example, the number 11111 shows that there are no problems in any of the 5 dimensions.
Evolution over time in the quality of life of patients in the "controls" group - EQ5D-5L | At the end of study visit, 2 months +/- 15 days after inclusion
  The EQ-5D (EuroQoL -5 Dimension) self-report questionnaire will be used to measure the quality of life under various health conditions and treatments according to 5 dimensions: mobility, personal autonomy, everyday living activities, pain/discomfort and anxiety/depression. There are 3 versions of this questionnaire: EQ-5D-3L with 3 levels of severity for each dimension, EQ-5D-5L with 5 levels of severity for each dimension and EQ-5D-Y which is the children's version. Each version is available in several languages. The questionnaire has 2 pages : page one with 5 items representing the 5 dimensions and page two with a visual analogue scale graded from 0 to 100 with 100 as the best possible state of health. For each dimension the patient must indicate what condition he/she is in. When all the answers are combined, a 5-figure number is obtained, indicating the patient's health condition. For example, the number 11111 shows that there are no problems in any of the 5 dimensions.
Side-effects related to immunotherapy in "cases" group - patient's viewpoint. | At the inclusion visit on Day 0
  The NCI PRO-CTCAE (National Cancer Institute - Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale will be used to evaluate the side-effects of treatment so that they can be declared for clinical studies in cancerology. The measurement of the result is declared directly by the patient based on the last seven days of treatment. The choice of terms and the categories of toxicity depend on the adverse events targeted. A French version is available on the following link: https://healthcaredelivery.cancer.gov/pro-ctcae/countries.html. The questionnaire for this particular study will be created on the PROCTCAE website via the option "build a custom form" (https://healthcaredelivery.cancer.gov/pro-ctcae/builder.html). 20 symptoms or side effects that may occur during treatment will be selected to build a patient-reported outcomes questionnaire adapted to the study.
Side-effects related to immunotherapy in "cases" group - patient's viewpoint. | At the follow-up visit, 1 month +/- 7 days after inclusion
  The NCI PRO-CTCAE (National Cancer Institute - Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale will be used to evaluate the side-effects of treatment so that they can be declared for clinical studies in cancerology. The measurement of the result is declared directly by the patient based on the last seven days of treatment. The choice of terms and the categories of toxicity depend on the adverse events targeted. A French version is available on the following link: https://healthcaredelivery.cancer.gov/pro-ctcae/countries.html. The questionnaire for this particular study will be created on the PROCTCAE website via the option "build a custom form" (https://healthcaredelivery.cancer.gov/pro-ctcae/builder.html). 20 symptoms or side effects that may occur during treatment will be selected to build a patient-reported outcomes questionnaire adapted to the study.
Side-effects related to immunotherapy in "cases" group - patient's viewpoint. | At the end of study visit, 2 months +/- 15 days after inclusion
  The NCI PRO-CTCAE (National Cancer Institute - Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale will be used to evaluate the side-effects of treatment so that they can be declared for clinical studies in cancerology. The measurement of the result is declared directly by the patient based on the last seven days of treatment. The choice of terms and the categories of toxicity depend on the adverse events targeted. A French version is available on the following link: https://healthcaredelivery.cancer.gov/pro-ctcae/countries.html. The questionnaire for this particular study will be created on the PROCTCAE website via the option "build a custom form" (https://healthcaredelivery.cancer.gov/pro-ctcae/builder.html). 20 symptoms or side effects that may occur during treatment will be selected to build a patient-reported outcomes questionnaire adapted to the study.
Side-effects related to immunotherapy in "controls" group - patient's viewpoint. | At the inclusion visit on Day 0
  The NCI PRO-CTCAE (National Cancer Institute - Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale will be used to evaluate the side-effects of treatment so that they can be declared for clinical studies in cancerology. The measurement of the result is declared directly by the patient based on the last seven days of treatment. The choice of terms and the categories of toxicity depend on the adverse events targeted. A French version is available on the following link: https://healthcaredelivery.cancer.gov/pro-ctcae/countries.html. The questionnaire for this particular study will be created on the PROCTCAE website via the option "build a custom form" (https://healthcaredelivery.cancer.gov/pro-ctcae/builder.html). 20 symptoms or side effects that may occur during treatment will be selected to build a patient-reported outcomes questionnaire adapted to the study.
Side-effects related to immunotherapy in "controls" group - patient's viewpoint. | At the follow-up visit, 1 month +/- 7 days after inclusion
  The NCI PRO-CTCAE (National Cancer Institute - Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale will be used to evaluate the side-effects of treatment so that they can be declared for clinical studies in cancerology. The measurement of the result is declared directly by the patient based on the last seven days of treatment. The choice of terms and the categories of toxicity depend on the adverse events targeted. A French version is available on the following link: https://healthcaredelivery.cancer.gov/pro-ctcae/countries.html. The questionnaire for this particular study will be created on the PROCTCAE website via the option "build a custom form" (https://healthcaredelivery.cancer.gov/pro-ctcae/builder.html). 20 symptoms or side effects that may occur during treatment will be selected to build a patient-reported outcomes questionnaire adapted to the study.
Side-effects related to immunotherapy in "controls" group - patient's viewpoint. | At the end of study visit, 2 months +/- 15 days after inclusion
  The NCI PRO-CTCAE (National Cancer Institute - Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale will be used to evaluate the side-effects of treatment so that they can be declared for clinical studies in cancerology. The measurement of the result is declared directly by the patient based on the last seven days of treatment. The choice of terms and the categories of toxicity depend on the adverse events targeted. A French version is available on the following link: https://healthcaredelivery.cancer.gov/pro-ctcae/countries.html. The questionnaire for this particular study will be created on the PROCTCAE website via the option "build a custom form" (https://healthcaredelivery.cancer.gov/pro-ctcae/builder.html). 20 symptoms or side effects that may occur during treatment will be selected to build a patient-reported outcomes questionnaire adapted to the study.
Side-effects related to immunotherapy in "cases" group - clinician's viewpoint. | At the inclusion visit on Day 0
  Version 4.03 of the NCI-CTCAE (National Cancer Institute- Common Terminology Criteria for Adverse Events) scale in French will be used to declare adverse events. It has 26 categories describing over 300 undesirable events, graded according to their severity (5 grades, each with its unique medical term). Grade 1 = Slight; asymptomatic or slight symptoms, only diagnosed upon clinical examination, requiring no treatment. Grade 2 = Moderate; requiring minimum local or non-invasive treatment; interfering with instrumental activities of daily living.Grade 3 = Severe or medically significant but vital prognosis is not compromised. Indication for hospitalisation or prolongation of hospitalisation, invalidating, interfering with simple activities of daily living. Grade 4 = vital prognosis compromised, requiring emergency management. Grade 5 = Death due to the adverse event. Not all grades are appropriate for all adverse events and therefore some are listed with a choice of below Grade 5.
Side-effects related to immunotherapy in "cases" group - clinician's viewpoint. | At the follow-up visit, 1 month +/- 7 days after inclusion
  Version 4.03 of the NCI-CTCAE (National Cancer Institute- Common Terminology Criteria for Adverse Events) scale in French will be used to declare adverse events. It has 26 categories describing over 300 undesirable events, graded according to their severity (5 grades, each with its unique medical term). Grade 1 = Slight; asymptomatic or slight symptoms, only diagnosed upon clinical examination, requiring no treatment. Grade 2 = Moderate; requiring minimum local or non-invasive treatment; interfering with instrumental activities of daily living.Grade 3 = Severe or medically significant but vital prognosis is not compromised. Indication for hospitalisation or prolongation of hospitalisation, invalidating, interfering with simple activities of daily living. Grade 4 = vital prognosis compromised, requiring emergency management. Grade 5 = Death due to the adverse event. Not all grades are appropriate for all adverse events and therefore some are listed with a choice of below Grade 5.
Side-effects related to immunotherapy in "cases" group - clinician's viewpoint. | At the end of study visit, 2 months +/- 15 days after inclusion
  Version 4.03 of the NCI-CTCAE (National Cancer Institute- Common Terminology Criteria for Adverse Events) scale in French will be used to declare adverse events. It has 26 categories describing over 300 undesirable events, graded according to their severity (5 grades, each with its unique medical term). Grade 1 = Slight; asymptomatic or slight symptoms, only diagnosed upon clinical examination, requiring no treatment. Grade 2 = Moderate; requiring minimum local or non-invasive treatment; interfering with instrumental activities of daily living.Grade 3 = Severe or medically significant but vital prognosis is not compromised. Indication for hospitalisation or prolongation of hospitalisation, invalidating, interfering with simple activities of daily living. Grade 4 = vital prognosis compromised, requiring emergency management. Grade 5 = Death due to the adverse event. Not all grades are appropriate for all adverse events and therefore some are listed with a choice of below Grade 5.
Side-effects related to immunotherapy in "controls" group - clinician's viewpoint. | At the inclusion visit on Day 0
  Version 4.03 of the NCI-CTCAE (National Cancer Institute- Common Terminology Criteria for Adverse Events) scale in French will be used to declare adverse events. It has 26 categories describing over 300 undesirable events, graded according to their severity (5 grades, each with its unique medical term). Grade 1 = Slight; asymptomatic or slight symptoms, only diagnosed upon clinical examination, requiring no treatment. Grade 2 = Moderate; requiring minimum local or non-invasive treatment; interfering with instrumental activities of daily living.Grade 3 = Severe or medically significant but vital prognosis is not compromised. Indication for hospitalisation or prolongation of hospitalisation, invalidating, interfering with simple activities of daily living. Grade 4 = vital prognosis compromised, requiring emergency management. Grade 5 = Death due to the adverse event. Not all grades are appropriate for all adverse events and therefore some are listed with a choice of below Grade 5.
Side-effects related to immunotherapy in "controls" group - clinician's viewpoint. | At the follow-up visit, 1 month +/- 7 days after inclusion
  Version 4.03 of the NCI-CTCAE (National Cancer Institute- Common Terminology Criteria for Adverse Events) scale in French will be used to declare adverse events. It has 26 categories describing over 300 undesirable events, graded according to their severity (5 grades, each with its unique medical term). Grade 1 = Slight; asymptomatic or slight symptoms, only diagnosed upon clinical examination, requiring no treatment. Grade 2 = Moderate; requiring minimum local or non-invasive treatment; interfering with instrumental activities of daily living.Grade 3 = Severe or medically significant but vital prognosis is not compromised. Indication for hospitalisation or prolongation of hospitalisation, invalidating, interfering with simple activities of daily living. Grade 4 = vital prognosis compromised, requiring emergency management. Grade 5 = Death due to the adverse event. Not all grades are appropriate for all adverse events and therefore some are listed with a choice of below Grade 5.
Side-effects related to immunotherapy in "controls" group - clinician's viewpoint. | At the end of study visit, 2 months +/- 15 days after inclusion
  Version 4.03 of the NCI-CTCAE (National Cancer Institute- Common Terminology Criteria for Adverse Events) scale in French will be used to declare adverse events. It has 26 categories describing over 300 undesirable events, graded according to their severity (5 grades, each with its unique medical term). Grade 1 = Slight; asymptomatic or slight symptoms, only diagnosed upon clinical examination, requiring no treatment. Grade 2 = Moderate; requiring minimum local or non-invasive treatment; interfering with instrumental activities of daily living.Grade 3 = Severe or medically significant but vital prognosis is not compromised. Indication for hospitalisation or prolongation of hospitalisation, invalidating, interfering with simple activities of daily living. Grade 4 = vital prognosis compromised, requiring emergency management. Grade 5 = Death due to the adverse event. Not all grades are appropriate for all adverse events and therefore some are listed with a choice of below Grade 5.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - ICM parc euromedecine, Montpellier, Hérault
  - Hopital Tenon ( Paris), Paris, Paris Cx 20
  - Institut Sainte Cancerologie Lucien Neuwirth, Avignon, Saint Priest En Jarez
  - ICO-Site Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - HEGP GH Universitaire Paris Ouest, Paris
  - ICANS Strasbourg, Strasbourg
  - Iuct Oncopole, Toulouse

REFERENCES:
- [Result] Annakib S, Fiteni F, Houede N. Quality of Life with Monoclonal Antibody Therapies for Locally Advanced or Metastatic Urothelial Carcinoma: A Systematic Review. Eur Urol Oncol. 2023 Oct;6(5):467-476. doi: 10.1016/j.euo.2023.05.001. Epub 2023 May 25. PMID 37244802
- [Derived] Annakib S, Di Meglio E, Dibert-Bekoy Y, Chevallier T, Roubaud G, Fournel P, Guillot A, Borchiellini D, Pouessel D, Boughalem E, Delva R, Barthelemy P, Oudard S, Thibault C, Tosi D, Houede N, Fiteni F. Patient Versus Clinician Reported Symptoms Agreement in Advanced Metastatic Bladder Cancer Patients. Cancer Med. 2025 Apr;14(8):e70896. doi: 10.1002/cam4.70896. PMID 40256972